CLINICAL TRIAL: NCT04609540
Title: Pyrotinib Combined With Trastuzumab and Chemotherapy in HER2-positive Metastatic Breast Cancer Patients- a Multicenter Retrospective Study
Brief Title: Pyrotinib Combined With Trastuzumab And Chemotherapy in HER2-positive MBC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Zhiyong Yu, Principal Investigator, Shandong Cancer Hospital and Institute
Other Study IDs: ShandongCHI-14
Record Dates: First submitted 2020-10-24; First posted 2020-10-30 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-10

CONDITIONS: HER2-positive Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pyrotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pyrotinib and Trastuzumab group: Dual anti-HER2 therapy (pyrotinib and trastuzumab) and chemotherapy
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Dual anti-HER2 therapy
  Other Names: Pyrotinib

SUMMARY:
To explore the real world data of trastuzumab Combined With Trastuzumab And Chemotherapy in China, and to explore the relationship between progression free survival and treatment pattern.

ELIGIBILITY:
Inclusion Criteria:

* woman, age > 18 years old
* Diagnosed with HER2 +Metastatic Breast Cancer
* Pyrotinib Combined With Trastuzumab And Chemotherapy for at least one cycle, starting from 2020.11.01-2021.10.31
* Available medical history

Exclusion Criteria:

* Incomplete medical history

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 positive Metastatic Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | 1 year
  The time from starting pyrotinib until disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival(OS) | 1 year
  The time from starting pyrotinib until death, regardless of cause.
Objective Response Rate(ORR) | 1 year
  The proportion of patients with complete response (CR) or partial response (PR)
Safety | 1 year
  Number of participants with adverse events which were collected at 6 and 18 months after the start of pyrotinib

IPD SHARING:
Plan to Share IPD: No